CLINICAL TRIAL: NCT00650975
Title: ThromboAblation in Acute Myocardial Infarction
Acronym: TAAMI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow enrollment rate.
Sponsor: KCRI (Other)
Collaborators: Spectranetics Corporation (Industry)
Responsible Party: William Kerker, Sr. Manager, Clinical Applications Research, Spectranetics Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D001747-01
Record Dates: First submitted 2008-03-26; First posted 2008-04-02 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: ST Elevation Acute Myocardial Infarction
Keywords: STEMI; Laser; Thrombus; Thrombectomy
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELCA (Active Comparator): Laser Thromboablation
  Interventions: Device: Laser Thromboablation
- PTCA (Active Comparator): PTCA (Direct Stenting)
  Interventions: Device: PTCA (Direct Stenting)

INTERVENTIONS:
Device: Laser Thromboablation — Laser Thromboablation using the Spectranetics CVX-300® excimer laser system
  Arms: ELCA
Device: PTCA (Direct Stenting) — Balloon predilatation or Direct Stenting using conventional techniques according to local standards and device specific instructions for use
  Other Names: PCI; Direct Stenting
  Arms: PTCA

SUMMARY:
1. Assess whether excimer laser coronary atherectomy (ELCA) before direct infarct-related artery (IRA) stenting results in improved reperfusion success in patients presenting with acute ST wave elevation myocardial infarction (STEMI) and angiographically evident thrombus.
2. Validate an ELCA technique for the treatment of STEMI, at high-volume centers experienced in the treatment of acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

Electrocardiographic inclusion criteria: (baseline 12-lead ECG recorded at 25 mm/second upon arrival at investigational center)

* STEMI within 12 hours of symptom onset, with ≥ 2 mm ST segment elevation in two or more leads and minimum ≥ 3 mm ST segment elevation in one lead.

Angiographic inclusion criteria after crossing with guidewire:

* IRA is a native coronary artery; and,
* Reference vessel diameter 2.5 - 4.0 mm; and,
* TIMI 0 or 1 flow with any TIMI thrombus grade; or,
* TIMI 2 or 3 flow with TIMI thrombus grade 3 or greater

Exclusion Criteria:

* Patient unwilling or unable to give informed consent
* Previous MI in the distribution of the current IRA
* Previous CABG
* Contraindications to PCI

  * allergy(s) to intended study medications
  * contraindicated for stent implantation
* Active bleeding or coagulopathy
* Patient in cardiogenic shock (<90mmHg SBP and/or requiring IABP or vasopressors)
* Known left ventricular ejection fraction (EF) <30%
* Fibrinolytic administered before PCI
* Renal insufficiency (creatinine >2.0mg/dl)
* Current vitamin K antagonist therapy or known INR >1.5
* Known thrombocytopenia - platelets <100,000 cell count
* Patient has Left Bundle Branch Block (LBBB) or pacemaker rhythm
* Known history of hemorrhagic stroke (CVA or TIA) <2 years before screening
* Known or suspected pregnancy
* Current cancer disease
* Comorbidity where survival is anticipated to be <1 year.
* No future patient cooperation expected
* Patient is participating in another clinical study
* Patient <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-03; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Myocardial Blush Grade 3 (MBG3) ST-Resolution MACE | 60 minutes - 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, MD, PhD, Principal Investigator — Department of Haemodynamics and Angiocardiography Medical College Jagiellonian University University Hospital in Krakow
Locations (5):
- Poland (5):
  - Gornoslaskie Centrum Medyczne 3rd Dept of Cardiology, Katowice
  - Jagiellonian University College of Medicine, Institute of Cardiology John Paul II Hospital, Krakow
  - Department of Haemodynamics and Angiocardiography Medical College Jagiellonian University University Hospital in Krakow, Krakow
  - University Hospital No. 1 1st Dept. of Cardiology, Poznan
  - Institute of Cardiology Hemodynamics dept., Cardiac Catheterization Laboratory, Warsaw